CLINICAL TRIAL: NCT02733341
Title: The Effect of Intravenous Cangrelor and Oral Ticagrelor on Platelets, the Microcirculation and Myocardial Damage in Patients Admitted With STEMI Treated by Primary Percutaneous Coronary Intervention: A Randomized Controlled Pilot Trial
Brief Title: The Effect of IV Cangrelor and Oral Ticagrelor Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Royal Wolverhampton Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015CAR77
Record Dates: First submitted 2016-04-05; First posted 2016-04-11 (Estimated); Results first posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Acute Coronary Syndrome (ACS); High On-treatment Platelet Reactivity (HTPR); Microvascular Obstruction (MVO); ST-segment Elevation Myocardial Infarction (STEMI); Thrombolysis in Myocardial Infarction (TIMI); Unstable Angina (UA)
Keywords: Adenosine Diphosphate; Cardiovascular Magnetic Resonance (CMR); Index of microvascular resistance (IMR); Vasodilator stimulated phosphoprotein phosphorylation (VASP); Pharmacodynamic; Antiplatelet; Myocardial Infarction (MI); Cangrelor; Ticagrelor; Coronary artery bypass graft (CABG); Primary percutaneous coronary intervention (PPCI)
MeSH Terms: conditions — Acute Coronary Syndrome; ST Elevation Myocardial Infarction; Angina, Unstable; Myocardial Infarction | interventions — cangrelor; Ticagrelor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oral Ticagrelor (Active Comparator): Patients in the oral Ticagrelor arm will receive Ticagrelor at a loading dose of 180mg followed by maintenance dose of 90mg twice daily for 12 months.
  Interventions: Drug: Ticagrelor
- Intravenous Cangrelor (Active Comparator): Patients in the intravenous Cangrelor arm will receive Cangrelor as an initial bolus dose given as per body weight followed by an intravenous infusion for no longer than three hours, they will then switch to oral Ticagrelor given at maintenance dose of 90mg twice daily for 12 months
  Interventions: Drug: Cangrelor

INTERVENTIONS:
Drug: Cangrelor
  Arms: Intravenous Cangrelor
Drug: Ticagrelor
  Arms: Oral Ticagrelor

SUMMARY:
Major heart attacks are caused by a number of factors, the two major of which are furring up of a coronary artery with atheroma and then sudden clot formation on this area leading to a blockage and interruption of blood flow. The clots that lead to heart attacks are largely made of clotting blood cells (platelets) that in health repair blood vessels and inhibit spontaneous bleeding. One of the main treatment strategies for heart attacks is to make these cells less "sticky". Aspirin is a main stay of anti-platelet treatment in the United Kingdom (UK) and in addition one of three other oral antiplatelet agents acting on the same platelet activation pathway (P2Y12 receptor) is licensed for use. When a patient is admitted with a major heart attack, they are treated with emergency primary percutaneous coronary intervention (PPCI) a technique where a wire and balloon are used to reopen the coronary artery and then usually a stent (a slotted metal tube) is placed to keep the artery open. Aspirin and one of the P2Y12 inhibitor agents are given to prevent further clots and all have been shown to reduce negative events following heart attacks and angioplasty with stent insertion. There are increasing data, including from our own institution, showing that in the setting of heart attacks, the oral P2Y12 inhibitors are poorly absorbed and have little effect at the time of most need, i.e. soon after dosing while the primary PCI is being performed.

All three current P2Y12 inhibitor agents are taken in tablet form immediately before the emergency PPCI procedure. It appears that in healthy stable patients these agents take at least 30 min to 2 hours to have an adequate effect. In heart attack patients the angioplasty procedure is usually performed well within this timescale. Furthermore, patients who are having a heart attack do not have normal drug absorption with blood being diverted away from the stomach and gut activity being suppressed by other drugs such as morphine.

In this current study, patients with major heart attacks will be given our standard oral agent, Ticagrelor, or the newer intravenous agent Cangrelor prior to PPCI.

DETAILED DESCRIPTION:
The success of modern treatment for ST-segment elevation myocardial infarction (STEMI) is dependent, in part, on the adequate suppression of platelet activity. Primary percutaneous coronary intervention (PPCI) for STEMI management has led to marked reductions in morbidity and mortality (1, 2). Aspirin is the mainstay anti-platelet agent. It is rapidly absorbed in the upper gastrointestinal (GI) tract and results in a measurable inhibition of platelet function within 60 minutes (3, 4). The advent of the platelet P2Y12 inhibitors has led to further improvement in outcomes in patients with acute coronary syndromes (ACS) undergoing PCI with reduced ischaemic complications (5) albeit at an increase in rate of bleeding complications. These agents have a synergistic effect on platelet function with the addition of Clopidogrel to Aspirin leading to approximately 20% reduction in negative cardiovascular events (6).

Activation of platelets leads to a conformational change in the surface glycoprotein IIb/IIIa receptor that allows cross bridging with fibrinogen and rapid aggregation (platelet thrombus formation) (7, 8) During PPCI, thrombus formation and dispersion can have a major impact on outcome. Intravenous platelet IIb/IIIa receptor antagonists such as Abciximab were initially shown to have a positive impact on primary angioplasty outcomes leading to a class IIa indication within the European Society of Cardiology (ESC) guidelines for use in the treatment of STEMI with angioplasty (9).

As oral antiplatelet inhibition has improved (specifically with the addition of Clopidogrel, Prasugrel or Ticagrelor) there has been a concomitant reduction in the use of intravenous IIb/IIIa agents during PCI for patients with ACS. This has been partly informed by later studies suggesting that the additive value of these agents to dual anti-platelet therapy is questionable (10).

In addition, the extra bleeding complications are seen by some to be excessive (11).

Current NICE recommendations for the treatment of STEMI include Aspirin plus one of the P2Y12 agents Clopidogrel, Prasugrel or Ticagrelor.

Ticagrelor, a reversible p2Y12 agent (cyclopentyltriazolopyrimidine CPTP) has been shown to be superior to Clopidogrel in ACS patients in the PLATO trial (12).

In this multicenter, randomized, double-blind trial, 18,624 patients were recruited. 7544 patients with STEMI were allocated to either Ticagrelor 180mg loading dose followed by 90 mg twice daily or Clopidogrel 300mg loading dose followed by 75 mg daily for 6 to 12 months. At 12 months, the primary end point - a composite of death from vascular causes, myocardial infarction, or stroke - had occurred in 9.8% of patients receiving Ticagrelor as compared with 11.7% of those receiving Clopidogrel (hazard ratio, 0.84; 95% confidence interval [CI], 0.77 to 0.92; P<0.001). Predefined hierarchical testing of secondary end points showed significant differences in the rates of other composite end points, as well as myocardial infarction alone (5.8% in the Ticagrelor group vs. 6.9% in the Clopidogrel group, P=0.005) and death from vascular causes (4.0% vs. 5.1%, P=0.001) but not stroke alone (1.5% vs. 1.3%, P=0.22). The rate of death from any cause was also reduced with Ticagrelor (4.5%, vs. 5.9% with Clopidogrel; P<0.001) (12)

We currently use Ticagrelor in patients admitted with STEMI prior to PPCI. Recently published data suggests however that even with this rapidly effective oral agent, it is not fully functional at the time of PPCI given the short timelines involved (13, 14)

Ticagrelor differs from the thienopyridine class of antiplatelet agents (Clopidogrel, Prasugrel, and Ticlopidine) as it does not exist as a prodrug and thus does not require biotransformation by hepatic enzymes before becoming active. Also Ticagrelor binds reversibly to P2Y12 receptors leading to a faster onset and offset than Clopidogrel (15).

Moreover, in the RESPOND study, Ticagrelor therapy was associated with uniform and superior platelet inhibition in both previously identified Clopidogrel responders and non-responders, and that inhibition, in turn, was associated with an extremely low prevalence of high on-treatment platelet reactivity (16).

Ticagrelor has recently received recommendation in the ESC guideline as a front-line treatment option for STEMI and NSTEMI (17, 18)

Ideally a full antiplatelet effect would be evident at the start of the PPCI, whereas in practice dosing of Clopidogrel, Prasugrel or Ticagrelor typically occurs on admission to hospital (possible only 10-20 minutes prior to PPCI).

Cangrelor is an adenosine diphosphate analogue that reversibly binds to and inhibits the P2Y12 ADP receptor. It has a half-life of 3 to 6 minutes and, when given as a bolus plus infusion, quickly and consistently inhibits platelets to a high degree, with normalisation of platelet function within 60 minutes after discontinuation (19).

Cangrelor [Kengrexal (EU), Kengreal (USA)] has been licensed for use in Europe, USA and the UK since March 2015, June 2015 and July 2015 respectively. Co-administered with Aspirin, is indicated for the reduction of thrombotic cardiovascular events in adult patients with coronary artery disease undergoing percutaneous coronary intervention (PCI) who have not received an oral P2Y12 inhibitor prior to the PCI procedure and in whom oral therapy with P2Y12 inhibitors is not feasible or desirable.

The use of Cangrelor in patients undergoing PCI has been studied in three phase 3 trials, the Cangrelor versus Standard Therapy to Achieve Optimal Management of Platelet Inhibition (CHAMPION) PCI study, the CHAMPION PLATFORM study and the CHAMPION PHOENIX study (19)(20)(21). In the CHAMPION PCI and the CHAMPION PLATFORM studies, Cangrelor, compared to oral Clopidogrel was not associated with a significant reduction in the primary efficacy end point (All cause death, MI or ischaemia driven revascularization at 48 hours) but was associated with reductions in secondary end points, including the rate of stent thrombosis, with no excess in severe bleeding. In the CHAMPION PLATFORM study there was also a reduction of the pre-specified secondary endpoint of death in the Cangrelor arm. The CHAMPION PHOENIX trial enrolled 11,145 patients undergoing PCI for SA, NSTEMI/UA or STEMI. Patients were randomized to either IV Cangrelor followed by Clopidogrel or oral Clopidogrel (300 or 600 mg) before during or immediately after PCI. In this study patients treated with the intravenous agent were significantly less likely to experience one of the primary endpoints (all cause death, MI or ischaemia driven revascularization at 48 hours), with no significant increase in bleeding. The study included 1992 patients with STEMI, who appeared to have a similar benefit to the SA and NSTEMI patients. Currently there are no data comparing the relative efficacy of Cangrelor with the more potent and rapidly acting Ticagrelor in patients undergoing PPCI for acute STEMI of less than 12 hours duration.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with STEMI eligible for PPCI
* Able to give verbal assent pre procedure and written consent following the procedure.
* Age ≥18 years
* No contraindication to Cangrelor or Ticagrelor
* Thienopyridine naïve

If a patient gives verbal assent but is unable to provide a written consent at a later stage due to incapacitation, presumed consent will be continued. The reasons why a patient becomes incapacitated and becomes unable to provide a written consent will be recorded during data collection.

Exclusion Criteria:

* Be unable to provide verbal assent and written consent
* Allergic to Aspirin or any of the P2Y12 antagonists in the trial
* Have pre-existing cardiogenic shock
* Previous myocardial infarction
* Have a concurrent septic or inflammatory disease e.g. rheumatoid arthritis, lupus, and pneumonia.
* Already taking a P2Y12 inhibitor
* Known bleeding diathesis
* Significant active bleeding
* History of intracranial hemorrhage
* Patients who are being treated with formal anticoagulation (Vitamin K antagonist, Factor II or Xa inhibitors) or have an indication for anticoagulation during the first four hours of the study period. Example is patients known to have atrial fibrillation, pulmonary embolism or deep vein thrombosis.
* Known severe renal dysfunction requiring renal replacement therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-07-21 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Cotton, Principal Investigator — The Royal Wolverhampton NHS Trust
Locations (1):
- The Royal Wolverhampton NHS Trust, Wolverhampton, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ubaid S, Ford TJ, Berry C, Murray HM, Wrigley B, Khan N, Thomas MR, Armesilla AL, Townend JN, Khogali SS, Munir S, Martins J, Hothi SS, McAlindon EJ, Cotton JM. Cangrelor versus Ticagrelor in Patients Treated with Primary Percutaneous Coronary Intervention: Impact on Platelet Activity, Myocardial Microvascular Function and Infarct Size: A Randomized Controlled Trial. Thromb Haemost. 2019 Jul;119(7):1171-1181. doi: 10.1055/s-0039-1688789. Epub 2019 May 26. PMID 31129911

RESULTS

PARTICIPANT FLOW:
Groups:
- Oral Ticagrelor: Patients in the oral Ticagrelor arm will receive Ticagrelor at a loading dose of 180mg followed by maintenance dose of 90mg twice daily for 12 months.
  Ticagrelor
- Intravenous Cangrelor: Patients in the intravenous Cangrelor arm will receive Cangrelor as an initial bolus dose given as per body weight followed by an intravenous infusion for no longer than three hours, they will then switch to oral Ticagrelor given at maintenance dose of 90mg twice daily for 12 months
  Cangrelor
Period: Overall Study
Arm/Group | Oral Ticagrelor | Intravenous Cangrelor
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients allocated to ticagrelor received a loading dose of 180mg of the drug orally immediately following randomization and prior to admission to the catheter suite. They then continued a maintenance dose of 90mg twice daily for 12 months as per standard clinical practice.
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Ticagrelor | Intravenous Cangrelor | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 31 | 27 | 58
  >=65 years | 19 | 23 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.4 (12.9) | 61.2 (13.9) | 62.3 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 11 | 28
  Male | 33 | 39 | 72
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Degree of Platelet Inhibition Measured
Description: P2Y12 inhibition was measured using VerifyNow™ rapid platelet function analyzer at the time of infarct vessel balloon inflation, 4 hours following study drug loading and at 24-36 hours. A single value was calculated by using the mean/average value.
  Results are expressed as P2Y12 reaction units (PRU), indicating the degree of ADP- mediated aggregation specific to the P2Y12 receptor. PRU values of ≥208 are indicative of a suboptimal response and are associated with poor clinical outcomes including death, MI and stroke at one year.
Time Frame: Measured at 4, 24 and 36 hours post dosing
Measure: Mean (Standard Deviation); unit: Platelet Reactivity Units (PRU)
Arm/Group | Oral Ticagrelor | Intravenous Cangrelor
Number analyzed (Participants) | 50 | 50
Platelet Reactivity Units (PRU) | 248.3 (55.1) | 145.2 (50.6)

2. Secondary Outcome: Index of Microvascular Resistance (IMR) Measurement
Description: Index of Microvascular Resistance (IMR) measurement using pressure wire studies immediately following the PPCI procedure.
  At the end of the clinical procedure a coronary pressure-/ temperature-sensitive guidewire (Radi Medical Systems, Uppsala, Sweden) will be utilised. The guidewire will be calibrated outside the body then equalized within the guide catheter, with the pressure sensor positioned at the ostium of the guide catheter. The guidewire microsensor will be advanced into the distal third of the culprit artery. The apparent IMR is calculated by multiplying the distal coronary pressure by the mean transit time of a 3 ml bolus of saline at room temperature during coronary hyperaemia induced by intravenous adenosine.
Time Frame: 1 hour
Measure: Mean (Standard Deviation); unit: mmHg*seconds
Arm/Group | Oral Ticagrelor | Intravenous Cangrelor
Number analyzed (Participants) | 50 | 50
mmHg*seconds | 131.2 (92.9) | 158.1 (92.1)

3. Secondary Outcome: Measurement of Thrombolysis in Myocardial Infarction (TIMI)
Description: Measurement of thrombolysis in myocardial infarction (TIMI) flow grade using TIMI Frame Count.
  The TFC is a simple, reproducible, objective, and quantitative index of coronary flow that allows standardization of TIMI flow grades and facilitates comparisons of angiographic end points between trials.
Time Frame: 3 Months
Measure: Mean (Standard Deviation); unit: frames per second
Arm/Group | Oral Ticagrelor | Intravenous Cangrelor
Number analyzed (Participants) | 50 | 50
frames per second | 60.1 (56.3) | 61.0 (50.0)

4. Secondary Outcome: ST Segment Resolution by ECG
Description: ST Segment Resolution by ECG at 90-120 minutes post PPCI
  A 12 lead EKG was recorded before coronary reperfusion and 90-120 minutes following PPCI to assess ST-segment resolution (STR). This variable was expressed as complete (>70%), incomplete (>30% to < 70%) or none (<30%).
Time Frame: 90-120 minutes post PPCI
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Ticagrelor | Intravenous Cangrelor
Number analyzed (Participants) | 50 | 50
Participants
  Complete | 36 | 32
  Partial | 7 | 11
  None | 7 | 7

5. Secondary Outcome: The Impact of Cangrelor vs Ticagrelor on Initial Myocardial Infarct Size Based on Peak Troponin
Description: High sensitivity cardiac troponin T (cTnT) was measured at 24-36 hours following PPCI
  A blood sample will be taken 24-36 hours post PPCI to determine peak high sensitivity troponin levels.
Time Frame: 24-36 hours
Measure: Median (Full Range); unit: nanograms per liter
Arm/Group | Oral Ticagrelor | Intravenous Cangrelor
Number analyzed (Participants) | 50 | 50
nanograms per liter | 55 [44.50 to 61.50] | 56.50 [47.50 to 59.25]

ADVERSE EVENTS:
Time Frame: 1 year
Description: All serious adverse events will be reported. Depending on the nature of the event the reporting procedures will be followed. Any questions concerning serious adverse events reporting will be directed to the Chief Investigator in the first instance. All serious adverse events will be reported to the appropriate regulatory and ethical authorities.
Arm/Group | Oral Ticagrelor | Intravenous Cangrelor
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 1/50
Other Adverse Events (participants affected / at risk) | 4/50 | 2/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Ticagrelor (N=50) | Intravenous Cangrelor (N=50)
Acute Pulmonary Oedema (Cardiac disorders) | 0 (0) | 1 (1) — Acute Pulmonary Oedema, needed CPAP/Intubation and Acute Ischemic MVR led to MVR Prosthetic + single graft to OM.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oral Ticagrelor (N=50) | Intravenous Cangrelor (N=50)
Hematoma (Blood and lymphatic system disorders) | 3 | 2
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-14): https://cdn.clinicaltrials.gov/large-docs/41/NCT02733341/Prot_SAP_000.pdf